CLINICAL TRIAL: NCT01081483
Title: A Blinded, Randomized, Placebo-controlled Phase 1 Study in Healthy Male Adults to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles of Single Doses of ABT-072
Brief Title: A Study of Single Doses of ABT-072 in Japanese Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry)
Responsible Party: Kazuhiko Sawa, Abbott Japan Co., Ltd
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-310
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C
Keywords: Healthy Volunteers; HCV Infections
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-072 Tablet (Active Comparator): ABT-072 50 mg Tablet, every day (QD), single ascending doses, groups 1-3
  Interventions: Drug: ABT-072
- Placebo (Placebo Comparator): Placebo Tablet, QD, single doses, groups 1-3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-072 — See arm description for more information
  Arms: ABT-072 Tablet
Drug: Placebo — See arm description for more information
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of blinded, single ascending oral doses of ABT 072 under non-fasting conditions in healthy adult Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy adult Japanese males

Exclusion Criteria:

* Use of any medications (prescription and over-the-counter), vitamins, or herbal supplements within the 2-week period prior to the first dose of study drug administration or within 10 half-lives of the respective medication, whichever is longer.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab).
* Positive screen for drugs of abuse, alcohol, or cotinine.
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessment | Day 1 to Day 4 and Day 15.
  Safety and tolerability assessment by the evaluation of vital signs, ECGs, physical exams, clinical lab testing and adverse event monitoring.
Pharmacokinetic profile evaluation | Day 1 to Day 4
  Single Dose Pharmacokinetic profile evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Kobayashi, Study Director — Abbott Japan Co.,Ltd
Locations (1):
- Kagoshima, Prefecture, Japan